CLINICAL TRIAL: NCT06739590
Title: Impact of Teacher-Student Interactive Immersive Mixed Reality (MR) Technology on the Effectiveness of Hepatobiliary Anatomy Education for Medical Students: A Randomized Clinical Trial
Brief Title: Effectiveness of Teacher-Student Interactive Immersive Mixed Reality Technology on Anatomy Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-KY-413-01
Record Dates: First submitted 2024-09-10; First posted 2024-12-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-08

CONDITIONS: Teaching Innovation; Medical Education; Anatomy Education
Keywords: Medical Education; Anatomy; Teaching Innovation; Surgeon Training; Mixed Reality
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Stratified Randomized Block Design
Who Masked: Participant
Masking Description: Participants remained unaware of the trial purpose and assessment metrics, only that they would be learning and practicing the anatomical structures and surgical planning of hepatobiliary surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control Group (Placebo Comparator): 21 participants were allocated to this group. They completed a background questionnaire and assessed their baseline emotions using the Medical Emotions Scale (MES) before commencing the study. Participants then took a pre-study test assessing their spatial knowledge of hepatobiliary anatomy and a surgical planning component, based on their assigned group. Following the learning process on a sample case, they retook the MES and subsequently completed a test on the designated test cases.
  Interventions: Behavioral: Learning with CT scans
- 3D Group (Experimental): 23 participants were allocated to this group. They completed a background questionnaire and assessed their baseline emotions using the MES prior to the study. They then completed a pre-study test focused on spatial knowledge of hepatobiliary anatomy and surgical planning. After engaging with the sample case, participants retook the MES and completed a test on the specified test cases.
  Intervention：Learning anatomical structures using three-dimensional visualization models displayed on a computer.
  Interventions: Behavioral: Learning with 3D visualization models
- MR Group (Experimental): 22 participants were allocated to this group. Participants completed a background questionnaire and assessed their baseline emotions using the MES before the study commenced. They participated in a training tutorial on utilizing the MR headset and completed a pre-study test evaluating spatial knowledge of hepatobiliary anatomy and surgical planning. After the learning process with the sample case, participants retook the MES, completed a test on the designated test cases, and filled out a post-use adverse reaction scale for the MR device.
  Intervention：Viewing and manipulating 3D visualization models to learn anatomical structures using the MR headset.
  Interventions: Radiation: Learning with 3D-MR visualization models

INTERVENTIONS:
Behavioral: Learning with CT scans — The average performance improvement in this group will serve as the baseline for learning achievable through conventional CT and MR imaging alone.
  Arms: Control Group
Behavioral: Learning with 3D visualization models — Learning anatomical structures using three-dimensional visualization models displayed on a computer.
  Arms: 3D Group
Radiation: Learning with 3D-MR visualization models — Viewing and manipulating 3D visualization models to learn anatomical structures using the MR headset.
  Arms: MR Group

SUMMARY:
Background:

Novice surgeons often struggle to translate anatomical knowledge into clinical practice, primarily due to a lack of resources, significant variability in anatomical structures, and limited hands-on experience. These challenges can lead to considerable deficiencies in clinical performance. Traditional educational methods, such as textbooks and CT imaging, frequently fall short in offering the depth necessary for effective application in surgical settings. Recent technological advancements, particularly in Augmented Reality (AR), Virtual Reality (VR), and Mixed Reality (MR), are revolutionizing surgical education by creating immersive learning environments. In complex fields like hepatobiliary surgery, the integration of MR allows for enhanced visualization of anatomical details, improving the understanding of vascular structures and tumor localization, which consequently boosts surgical training outcomes. However, most research to date has analyzed these technologies in isolation, with few studies investigating their collaborative benefits or effective integration into educational curricula.

This study aims to evaluate cognitive learning outcomes related to anatomical structures by employing various modalities, including traditional medical imaging, 3D models, and 3D-MR. Through cross-comparative analyses, investigators will assess the correlation between test scores and actual clinical performance, thereby gauging the impact of these modalities on the comprehension of intricate anatomical structures and their spatial visualization skills. Ultimately, this study aspire to develop a comprehensive anatomical teaching program that incorporates MR and 3D models to demonstrate the feasibility and efficacy of these innovative technologies in teaching liver and gallbladder anatomy.

Research Objectives: To compare the effectiveness of learning outcomes in anatomical structure learning between MR 3D modelling and general medical imaging, and to investigate which modalities lead to higher anatomical learning outcomes (primary outcome).

Hypothesis: Compared to plain images, 3D models of MR simulators can significantly improve learning performance, achieve better learning outcomes

DETAILED DESCRIPTION:
Background:

Effective surgical planning in hepatobiliary surgery requires a deep understanding of complex anatomical structures, fraught with variations and anomalies. Mastery of the intricate spatial relationships among these structures poses considerable challenges, especially for novice surgeons striving to acquire essential skills. Traditional educational materials, including textbooks and CT images, often lack the necessary depth for effective application. As a result, many novice surgeons face difficulties in translating anatomical knowledge into clinical practice during preoperative planning. Additionally, a scarcity of hands-on experience in real surgical environments exacerbates these issues, creating knowledge gaps that may compromise clinical performance.

Fortunately, advancements in technology are paving the way for improved surgical education. Augmented Reality (AR), Virtual Reality (VR), and Mixed Reality (MR) have emerged as revolutionary tools in this arena, particularly for distance learning. Recent innovations have fostered immersive learning environments that enhance the educational experience for both surgical educators and students. The integration of these immersive technologies with 3D modeling holds significant potential for medical anatomy education. Research indicates that transforming 2D images into 3D VR models significantly enhances the intuitive understanding of anatomical structures. Compared to traditional educational methods, this approach improves knowledge retention and supports more effective memory formation.

In the realm of hepatobiliary surgery, which involves intricate vascular and anatomical features, there is increasing focus on utilizing immersive technologies. MR technology allows for enhanced visualization of liver anatomy, improving the understanding of vascular structures and tumor localization, ultimately benefiting surgical training. VR technology provides real-time interaction with 3D simulated environments, making it a critical tool for advancing surgical knowledge and skills. Meanwhile, AR enhances the educational experience, while MR and VR collectively facilitate a comprehensive visualization of the complex structures of liver.

Purpose of the Study:

Despite the potential benefits of integrating these technologies into clinical practice, existing studies primarily utilize 3D or 3D-VR technologies in isolation, often comparing them only to traditional methods. Few investigations address the combined effects of these modalities, leading to inconsistent integration into training programs and challenging learning curves for novice surgeons. Additionally, the absence of robust quantitative assessment tools limits the theoretical support for these educational methodologies.

Consequently, this study aims to establish a framework for teaching anatomy that incorporates MR and 3D models. The research will assess the influence of these innovative technologies on comprehension of intricate anatomical structures and their spatial visualization abilities regarding three-dimensional forms. Ultimately, our goal is to confirm the feasibility and effectiveness of integrating these advanced technologies into hepatobiliary anatomy education.

Research Goals:

Evaluate cognitive learning outcomes related to anatomical structures using diverse learning modalities, including traditional medical imaging, 3D modeling, and 3D-MR.

Test the effectiveness of different modalities in learning hepatobiliary anatomical structures through cross-comparisons, verifying the correlation between scores and actual performance.

Design:

This is a three-arm, partially blinded, randomized controlled trial comparing the learning outcomes associated with 3D models and 3D-MR for teaching hepatic and gallbladder anatomy.

Participants: Medical students who meet the inclusion and exclusion criteria and have no prior experience interpreting hepatobiliary surgical imaging.

Tasks: Experts will issue relevant test questions on hepatobiliary surgery anatomy, and learning outcomes across different modalities will be evaluated based on test scores.

Intervention: A randomized allocation method will divide participants into a control group and a new technology group. The three groups will receive instruction on the anatomy of the hepatobiliary system through different methodologies.

1. Control group: Engages with routine CT and MR imaging for anatomical structure learning.
2. New technology group:

3D group: Learns anatomical structures using 2D and 3D models in a computer environment.

MR group: Engages in anatomical structure learning utilizing 3D models within an MR simulator.

ELIGIBILITY:
Inclusion Criteria:

* Full-time undergraduate clinical medicine students
* Postgraduate and trainees from accredited residency programs.

Exclusion Criteria:

* Participants who had previously used the new technology or similar simulators
* Participants lacking clinical anatomy learning experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2024-12-21 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Anatomical knowledge | Before and after the completion of the learning process, an average of 1 day
  Anatomists create relevant test questions and assess performance of participants; by comparing the results of baseline and post-study score of the Anatomy and Surgical Competence Test. The improvement in test scores serves as an indicator for evaluating learning outcomes.

SECONDARY OUTCOMES:
Differences in Emotional Intensity | Before and after the completion of the learning process, an average of 1 day
  Participants independently completed the Medical Emotions Scale (MES) both before and after the learning process to assess the intensity of their emotions.
  The Medical Emotions Scale consists of twenty-two single-item adjectives designed to assess state emotions across four categories: basic, achievement, epistemic, and social emotions. These emotions are organized into five sub-scales based on their valence (pleasant or unpleasant) and activation (level of physiological arousal): (1) positive activating, (2) positive deactivating, (3) negative activating, (4) negative deactivating, and (5) neutral. Each emotion is scored according to its intensity, with higher scores indicating a greater intensity or strength of the emotion.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from primary and secondary outcomes may be shared if other researchers have an interest in this data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2025-January 2026
Access Criteria: Researchers wanting access to the data will need to contact the principal investigator of the trial. Dr. Jian Yang.

REFERENCES:
- [Background] Balci D, Kirimker EO, Raptis DA, Gao Y, Kow AWC. Uses of a dedicated 3D reconstruction software with augmented and mixed reality in planning and performing advanced liver surgery and living donor liver transplantation (with videos). Hepatobiliary Pancreat Dis Int. 2022 Oct;21(5):455-461. doi: 10.1016/j.hbpd.2022.09.001. Epub 2022 Sep 8. PMID 36123242
- [Background] Moro C, Stromberga Z, Raikos A, Stirling A. The effectiveness of virtual and augmented reality in health sciences and medical anatomy. Anat Sci Educ. 2017 Nov;10(6):549-559. doi: 10.1002/ase.1696. Epub 2017 Apr 17. PMID 28419750
- [Background] Mateen M, Kan CYP. Education during COVID-19: Ready, headset, go! Clin Teach. 2021 Feb;18(1):90-91. doi: 10.1111/tct.13266. Epub 2020 Oct 2. No abstract available. PMID 33006439
- [Background] Kolla S, Elgawly M, Gaughan JP, Goldman E. Medical Student Perception of a Virtual Reality Training Module for Anatomy Education. Med Sci Educ. 2020 Jun 9;30(3):1201-1210. doi: 10.1007/s40670-020-00993-2. eCollection 2020 Sep. PMID 34457783
- [Background] Alharbi Y, Al-Mansour M, Al-Saffar R, Garman A, Alraddadi A. Three-dimensional Virtual Reality as an Innovative Teaching and Learning Tool for Human Anatomy Courses in Medical Education: A Mixed Methods Study. Cureus. 2020 Feb 24;12(2):e7085. doi: 10.7759/cureus.7085. PMID 32226686
- [Background] Ammanuel S, Brown I, Uribe J, Rehani B. Creating 3D models from Radiologic Images for Virtual Reality Medical Education Modules. J Med Syst. 2019 May 3;43(6):166. doi: 10.1007/s10916-019-1308-3. PMID 31053902